CLINICAL TRIAL: NCT00618696
Title: MT2005-13R - Phase I Open Label, Single Arm, Dose Escalation Trial to Evaluate the Biodistribution and Safety of AHN-12 in Patients With Advanced Leukemia
Brief Title: Yttrium Y 90 Anti-CD45 Monoclonal Antibody AHN-12 in Treating Patients With Advanced Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced with another study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Linda Burns, M.D., Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS039; UMN-MT2005-13R (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Blast Crisis; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AHN-12 (Experimental): 2.0, 5.0, 7.5, 10.0 or 12.5 mCi/m^2 of ^90Y-AHN-12 at Day 7/8
  Interventions: Biological: anti-CD45 monoclonal antibody AHN-12; Radiation: yttrium Y 90 anti-CD45 monoclonal antibody AHN-12

INTERVENTIONS:
Biological: anti-CD45 monoclonal antibody AHN-12 — 150 mg/m^2 cold antibody at Day 0
  Other Names: ^111In-AHN-12
Radiation: yttrium Y 90 anti-CD45 monoclonal antibody AHN-12 — Dose per scheduled level; 2.5-12.5 mCi/m^2
  Other Names: ^90Y-AHN-12

SUMMARY:
RATIONALE: Monoclonal antibodies can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Radioactive monoclonal antibodies, such as yttrium Y 90 monoclonal antibody, can find cancer cells and either kill them or carry cancer-killing substances to them without harming normal cells.

PURPOSE: This phase I trial is studying the side effects and best dose of a yttrium Y 90 monoclonal antibody and how much radiation is taken in by the organs in the body in treating patients with advanced leukemia or other hematologic disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish that a dose of 150 mg/m² of nonradiolabeled anti-CD45 monoclonal antibody AHN-12 results in normal biodistribution, normal-organ estimated radiation-absorbed dose of less than 20 Gy, and estimated radiation-absorbed dose of no more than 13 Gy to the red marrow.

Secondary

* To determine the maximum tolerated dose of yttrium Y 90 anti-CD45 monoclonal antibody AHN-12 (^90Y-AHN-12).
* To determine the human anti-mouse antibody (HAMA) response.
* To define, preliminarily, the antitumor activity of ^90Y-AHN-12.

OUTLINE: This is a dose-escalation study of yttrium Y 90 anti-CD45 monoclonal antibody AHN-12 (^90Y-AHN-12).

* Biodistribution: Patients receive nonradiolabeled monoclonal antibody AHN-12 IV and an imaging dose of indium Y 111 monoclonal antibody AHN-12 (^111In-AHN-12) IV over 10 minutes on day 0. Patients undergo whole-body gamma-camera imaging immediately following infusion, at 4-6 hours, and on days 1, 3, 4, and 7. Blood samples are collected prior to each imaging for dosimetry calculations and pharmacokinetics.

Patients also undergo bone marrow biopsy 16-24 hours after infusion for dosimetry calculations. Patients with the expected biodistribution of ^111In-AHN-12, an estimated radiation-absorbed dose to the normal organ of < 20 Gy, an estimated radiation-absorbed dose to the red marrow of ≤ 13 Gy, and a negative human anti-mouse antibody at day 7 proceed to the therapy portion.

* Treatment: Patients receive nonradiolabeled anti-CD45 monoclonal antibody AHN-12 IV over 60 minutes and escalating therapy doses of yttrium Y 90 anti-CD45 monoclonal antibody AHN-12 (^90Y-AHN-12) IV over 10 minutes on day 7 or 8.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD45+ diseases:

  * Acute lymphoblastic leukemia or acute myeloid leukemia (AML), meeting any of the following criteria:

    * Primary refractory disease
    * Relapsed disease, defined as persistent disease following a minimum of 2 different standard chemotherapy induction attempts at time of diagnosis or at relapse
  * Acute myelogenous leukemia (AML), primary refractory or relapsed disease - defined as persistent disease after a minimum of two different standard chemotherapy induction attempts at time of diagnosis or relapse
  * Advanced myelodysplastic syndrome (MDS) defined as > or = 15% bone marrow blasts following a minimum of one standard chemotherapy induction attempt
  * AML arising from preexisting MDS, refractory - defined as persistent disease following a minimum of one standard chemotherapy induction attempt
  * Chronic myelogenous leukemia (CML) following blast crisis (> or = 15% marrow blasts following a minimum of one standard chemotherapy induction attempt
* Peripheral leukemic blasts (by morphology) must be < 5,000/μL (hydroxyurea to control peripheral blast count allowed)
* Must have source of allogeneic stem cells (sibling, unrelated cord[s], or donor) identified prior to initiation of protocol therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Total bilirubin ≤ 2.5 times upper limit of normal (ULN)
* aspartate aminotransferase (AST) and Alanine transaminase (ALT) ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.3 mg/dL OR creatinine clearance ≥ 60 mL/min
* Left ventricular ejection fraction (LVEF) ≥ 45% by Multi Gated Acquisition Scan (MUGA) or echocardiogram (ECHO)
* Carbon Monoxide Diffusing Capacity (DLCO) (corrected) ≥ 50% of predicted
* Human anti-mouse antibody (HAMA) must be negative
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Human immunodeficiency virus (HIV) negative
* Recovered from all prior therapy
* At least 7 days since prior biologic agents

Exclusion Criteria:

* Bone marrow cellularity < 15%
* Known brain metastases or active central nervous system (CNS) disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ^90Y-AHN-12 or other agents used in study
* Uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic or congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* Other concurrent investigational agents
* Prior allogeneic transplantation
* Less than 60 days since prior autologous transplantation with relapsed disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Biodistribution of nonradiolabeled anti-CD45 monoclonal antibody AHN-12 | Within 1 hour, 4-6 hours, Days 1, 3, 4 and 7 post infusion

SECONDARY OUTCOMES:
Maximum tolerated dose of yttrium Y 90 anti-CD45 monoclonal antibody AHN-12 | Week 8
Presence of human antibody to murine antibody | at baseline and at 28 days, 90 days, and 6 months after completion of study treatment
Dose-limiting toxicity and response | at days 28 and 90 after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Burns, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States